CLINICAL TRIAL: NCT01949870
Title: A Phase I, Open-Label, Multi-Center Study to Assess the Safety and Tolerability of Selumetinib (AZD6244, ARRY-142886) in Combination With Cisplatin/Gemcitabine in Japanese Patients With Inoperable Locally Advanced or Metastatic Biliary Tract Cancer (BTC)
Brief Title: Selumetinib (AZD6244, ARRY-142886) J-BTC Phase 1 Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: change in the development strategy
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00075
Record Dates: First submitted 2013-09-10; First posted 2013-09-25 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Inoperable Locally Advanced or Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cisplatin; Gemcitabine; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selumetinib (Other): 25mg/day, 50mg/day and 75mg/day
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Selumetinib

INTERVENTIONS:
Drug: Cisplatin — day1 and day8 at each cycle
Drug: Gemcitabine — day1 and day8 at each cycle
Drug: Selumetinib — 25mg/day, 50mg/day and 75mg/day
  Other Names: AZD6244

SUMMARY:
The objective of this study is to investigate the safety and tolerability of oral dose of selumetinib in combination with chemotherapies (cisplatin and gemcitabine) in Japanese patients with advanced biliary tract cancer (BTC). In addition, the pharmacokinetic (PK) profile of selumetinib and chemotherapies will be investigated. Also, the Maximum tolerated dose (MTD) of selumetinib in combination with chemotherapies for Japanese BTC patients will be identified, if possible.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Patients must be ≥ 20 years
3. Histological or cytological confirmation of locally advanced or metastatic BTC (intra- or extra-hepatic, gallbladder or ampullary carcinoma)
4. Patients who are eligible for treatment with standard dose of cisplatin/gemcitabine combination regimen
5. World Health Organisation (WHO) performance status (PS) 0-1
6. Evidence of post-menopausal status or negative urine/serum pregnancy test for nonmenopausal female patients Women will be considered postmenopausal if they are amenorrheic for 1 year or more without an alternative medical cause. The following age-specific requirements apply: i) Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 1 year or more following cessation of exogenous hormonal treatments and with Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range.

ii) Women over 50 years old would be consider postmenopausal if they have been amenorrheic for 1 year or more following cessation of all exogenous hormonal treatments, radiation-induced oophorectomy with last menses > 1 year ago, chemotherapy-induced menopause with >1 year interval since last menses. Or surgical sterilisation (bilateral oophorectomy or hysterectomy). 7. Male patients should be willing to use barrier contraception for a specified period 8. A lesion that can be accurately assessed at baseline by CT or magnetic resonance imaging (MRI) and is suitable for repeated assessment in accordance with RECIST 9. Patients must have a life expectancy ≥16 weeks 10. Patients who can remain in Hospital from Cycle 0 Day 1 up to at least the completion of Cycle 1 Day 9 11. Patient is willing to provide fresh or archival tumour sample and biomarker blood sample.

-

Exclusion Criteria:

1. Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
   * Any investigational agents or study drugs from a previous clinical study within 4 weeks of the first dose of study treatment
   * Chemotherapy, immunotherapy or anticancer agents within 3 weeks of the first dose of study treatment
   * selumetinib(therefore, patients who have already participated in this study and been taken selumetinib) or any other MEK(Mitogen-activated protein kinase kinase or Mitogen-activated protein kinase (MAPK) / Extracellular signal-regulated kinase (ERK) kinase) 1/2 inhibitor in past
   * Cisplatin or gemcitabine in past
   * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
   * Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment
2. With the exception of alopecia, any unresolved toxicities from prior therapy ≥Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
3. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
4. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, such as,

   * active bleeding diatheses
   * active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
   * severe renal impairment, uncontrolled diabetes or renal transplant
   * acute uncontrolled infection
   * current unstable or uncompensated respiratory or cardiac disease
   * peripheral vascular disease including diabetic vasculopathy Screening for chronic conditions is not required
5. Any of the following cardiac criteria:

   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events (eg, heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or mean resting corrected QT interval (QTc) > 470 msec)
   * Uncontrolled hypertension (BP≥150/95 mmHg despite medical therapy)
   * Acute coronary syndrome within 6 months prior to starting treatment
   * Angina Canadian Cardiovascular Society Grade II-IV (despite medical therapy)
   * Symptomatic heart failure (NYHA [New York Heart Association ] II-IV)
   * Prior or current cardiomyopathy
   * Baseline left ventricular ejection fraction (LVEF) <55% measured by echocardiography or Multiple Gated Acquisition Scan (MUGA)
   * Atrial fibrillation with a ventricular rate >100 bpm at rest
   * Severe valvular heart disease
6. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count < 1.5 x 109/L
   * Platelet count < 100 x 109/L
   * Haemoglobin < 90 g/L
   * Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) > 2.5 times ULN
   * Total bilirubin > 1.5 times ULN
   * Creatinine clearance < 50 mL/min (measured or calculated by Cockcroft and Gault equation)
7. Any of the following ophthalmological criteria:

   * Current or past history of central serous retinopathy or retinal vein occlusion
   * Intraocular pressure >21 mmHg
   * Uncontrolled glaucoma (irrespective of intraocular pressure)
8. Inadequate biliary drainage
9. Symptomatic patients with interstitial pneumonitis or lung fibrosis confirmed by plain chest X-ray or chest CT
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of selumetinib
11. History of hypersensitivity to selumetinib or drugs with a similar chemical structure or class to selumetinib
12. History of hypersensitivity to platinum and gemcitabine containing drugs
13. Use of strong CYP(Cytochrome P450)1A2, CYP(Cytochrome P450)2C19 or CYP3A4 inducers and/or inhibitors (for example, but not limited to, fluvoxamine, fluconazole, ticlopidine, ketoconazole, atazanavir, clarithromycin, indinavir, itraconazole, nelfinavir, ritonavir, saquinavir,telithromycin, voriconazole, grapefruit and seville orange or the juices of these fruits, rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort)
14. Any contraindication to the combination chemotherapy as per local prescribing information
15. Judgment by the investigators that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
16. Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site).

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - AZD6244 PhI Japanese Gem/, Kashiwa Shi, Chiba
  - AZD6244 PhI Japanese Gem/, Chuo Ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 study centres in Japan between October 2013 and August 2014.
Groups:
- Selumetinib+ Cisplatin + Gemcitabine: Selumetinib (25 mg bd)
  For each 21-day cycle:
  Cisplatin (25 mg/m2) Days 1 and 8 Gemcitabine (1000 mg/m2) Days 1 and 8
Period: Overall Study
Arm/Group | Selumetinib+ Cisplatin + Gemcitabine
Started | 6
Received Treatment | 4
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1
Not completed — Study termination | 1
Not completed — Eligibility requirements not fulfilled | 2

BASELINE CHARACTERISTICS:
Arm/Group | Selumetinib+ Cisplatin + Gemcitabine
Number analyzed (Participants) | 4
Age, Customized [Number; unit: Participants]
  <50 years | 1
  >=50 to < 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Dose-limiting Toxicities
Description: The number of dose-limiting toxicities in selumetinib in combination with cisplatin and gemcitabine
Time Frame: The first cycle with selumetinib until Day 1 of Cycle 2 of combination dosing
Population: Evaluable = completed at least 75% of planned daily doses of selumetinib at least 50% of planned dose of cisplatin/gemcitabine planned on Cycle 1 Day 8 (therefore, in total with Cycle 1 Day 1, at least 75 % of planned dose is given in Cycle 1) and has enough information to be assessed for the combination regimen dose escalation.
Measure: Number; unit: Participants
Arm/Group | Selumetinib+ Cisplatin + Gemcitabine
Number analyzed (Participants) | 3
Participants
  Yes | 0
  No | 3

ADVERSE EVENTS:
Time Frame: AEs were collected throughout the study, from informed consent until the end of the followup period (28 days after last dose).
Arm/Group | Selumetinib+ Cisplatin + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib+ Cisplatin + Gemcitabine (N=4)
Cholangitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib+ Cisplatin + Gemcitabine (N=4)
Anaemia (Blood and lymphatic system disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Oedema (General disorders) | 1
Platelet count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1

LIMITATIONS AND CAVEATS:
Dose escalation stopped after the first cohort due to changes in the drug development strategy. As such, a non-tolerated dose was not determined and the maximum tolerated dose could not be confirmed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less